CLINICAL TRIAL: NCT03487367
Title: Clinical Trial Readiness for SCA1 and SCA3
Acronym: READISCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: University of Michigan (Other); University of Minnesota (Other); University of Utah (Other); University of California, Los Angeles (Other); University of Chicago (Other); University of South Florida (Other); Harvard University (Other); Johns Hopkins University (Other); University of Florida (Other); Columbia University (Other); Emory University (Other); University of California, San Francisco (Other); University of Alabama at Birmingham (Other); University of Colorado, Denver (Other); University of Rochester (Other); Stanford University (Other); Northwestern University (Other); German Center for Neurodegenerative Diseases (DZNE) (Other); Institut de Recherche sur la Moelle épinière et l'Encéphale (Other); University of Pennsylvania (Other); Ohio State University (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, Tetsuo Ashizawa, MD, HMRI Neurosciences Principal Investigator & Multicenter Lead Investigator, The Methodist Hospital Research Institute
Other Study IDs: Pro00017836; U01 - Ashizawa 2016 (Other: HMRI)
Record Dates: First submitted 2018-03-01; First posted 2018-04-04 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia 3
Keywords: spinocerebellar ataxia; ataxia; ataxias; SCA1; SCA3; spinocerebellar ataxia type 1; spinocerebellar ataxia type 3; READISCA; SCA; SCAs; clinical trial readiness
MeSH Terms: conditions — Spinocerebellar Ataxias; Machado-Joseph Disease; Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood collected for DNA analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early stage subjects: This cohort is defined by individuals with a total SARA score of less than or equal to 9.5
- Premanifest mutation carriers: This cohort is defined by the presence of positive genetic diagnosis but no signs of ataxia and total SARA score of less than or equal to 2.5
- 50%-at-risk subjects: This cohort is defined by individuals who are at risk for SCA1 or SCA3 because they have a family member who tested positive for SCA1 or SCA3. Total SARA score is less than or equal to 2.5
- Previously diagnosed early stage: This cohort is defined by individuals who were included in prior CRC-SCA, EUROSCA, ESMI or SPATAX studies who had a total SARA score of less than or equal to 10 in 2009-2012

SUMMARY:
The investigators plan to fill the gap between the current state of clinical trial readiness and the optimal one for SCA1 and SCA3, which are fatal rare diseases with no treatments. Through US-European collaborations, the investigators will establish the world's largest cohorts of subjects at the earliest disease stages, who will benefit most from treatments, validate an ability to detect disease onset and early progression by imaging markers, even prior to ataxia onset, and identify clinical trial designs that will generate the most conclusive results on treatment efficacy with small populations of patients.

DETAILED DESCRIPTION:
Spinocerebellar ataxia types 1 (SCA1) and 3 (SCA3) are rare, inherited neurodegenerative disorders that relentlessly progress to total disability and death. SCA1 is the fastest progressing SCA while SCA3 is the most common SCA in US and Europe. Expanded (CAG)n repeats encoding polyglutamines (polyQ) in the respective genes, Ataxin 1 (ATXN1) and Ataxin 3 (ATXN3), cause SCA1 and SCA3. Disease-modifying therapies that target the pathway upstream of the complex pathogenic cascade will offer ultimate treatment. Scientific premise and preclinical animal data strongly support MSK1 inhibitors for SCA1, citalopram for SCA3, and nucleotide-based gene silencing for both SCAs as drugs to be examined in clinical trials in five years. However, the challenge that investigators face in current clinical trial readiness for such disease-modifying therapies is that the modest effect size of candidate drugs as measured by the Scale for the Assessment and Rating of Ataxia (SARA; the most robust and well-validated clinical outcome assessment measure) requires large cohorts of study subjects to achieve sufficient statistical power. To accomplish the goal of establishing clinical trial readiness, the investigators propose to launch an international, multi-site effort focusing on premanifest mutation carriers and patients in an early disease stage, who are likely responders to the disease-modifying interventions prior to irreversible brain damage. Based on the investigators' studies funded by NIH and the National Ataxia Foundation (NAF), the US ataxia consortium has developed an unprecedented opportunity for tight collaborations with the European Ataxia Study Group to jointly address this challenge and establish clinical trial readiness for SCA1 and SCA3. To achieve this goal, the investigators propose the following specific aims:

Aim 1. Establish the world's largest cohorts of premanifest/early SCA1 and SCA3 by combining cohorts, clinical outcome assessment data and biofluid samples (blood, cerebrospinal fluid) from US and Europe Aim 2. Validate MR morphological, biochemical and functional biomarkers in premanifest and early SCA1 and SCA3 Aim 3. Adapt recent developments on statistical design and analysis of small population trials to SCAs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (no study-related procedures may be performed before the subject has signed the consent form).
2. Subjects of either sex aged 18 to 65 with presence of symptomatic ataxic disease or asymptomatic mutation carrier or
3. Subjects with definite molecular diagnosis of SCA1 or SCA3 or another affected family member
4. Subjects of any age with previous diagnosis of Early stage SCA1 and SCA3
5. Subjects capable of understanding and complying with protocol requirements
6. No changes in physical/occupational therapy status within two months prior to enrollment

Exclusion Criteria:

1. Subjects currently receiving, or having received within 2 months prior to enrollment into this study, any investigational drug.
2. Subjects who do not wish to or cannot comply with study procedures.
3. Genotype consistent with other inherited ataxias
4. Changes in coordinative physical and occupational therapy for ataxia 2 months prior to study participation
5. Concomitant disorder(s) or condition(s) that affects assessment of ataxia or severity of ataxia during this study
6. AIM 2 exclusion criteria also includes the inability to undergo MRI scanning and weight over 300lbs, presence of structural abnormalities such as subdural hematoma or primary or metastatic neoplasms and concurrent illnesses or treatment interfering with cognitive function such as stroke or normal pressure hydrocephalus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Early stage subjects refer to individuals who tested positive for the SCA1 or SCA3 gene mutation but show signs of ataxia
  2. Premanifest mutation carriers refer to individuals who who tested positive for the SCA1 or SCA3 gene mutation but do not show signs of ataxia
  3. 50%-at-Risk subjects refer to individuals who are at risk for developing SCA1 or SCA3 because they have an affected family member who tested positive for the gene mutation.
  4. Previously diagnosed early stage patients refer to individuals who previously participated between 2009-2012 in the CRC-SCA, ESMI, EUROSCA, or SPATAX studies. At time of previous participation total SARA score must be less than or equal to 10.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in disease progression in SCA1 and SCA3 as determined by change in scale for the assessment and rating of ataxia (SARA) score over time. | Every 12 months for approximately 60 months
  Scale for the assessment and rating of ataxia (SARA) was evaluated in two large validation trials performed by the EUROSCA clinical group and was found to be easy to use, reliable and valid. SARA has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
Change in disease progression in SCA1 and SCA3 as determined by change in Composite Cerebellar Functional Severity Score (CCFS) total score over time. | Every 12 months for approximately 60 months
  Composite Cerebellar Functional Severity Score (CCFS) is a validated quantitative scale used to evaluate cerebellar ataxia in adults and children. Total score calculation includes both the 9-hole pegboard test and the click test. A higher score indicates more severe cerebellar impairment.
Change in disease progression in SCA1 and SCA3 as determined by change in timed 25 foot walk test (T25FW) over time. | Every 12 months for approximately 60 months
  Timed 25 foot walk test (T25FW) is a quantitative mobility and leg function performance test based on a timed 25-walk. The T25FW has high inter-rater and test-retest reliability and shows evidence of good concurrent validity. Gait speed in general has been demonstrated to be a useful and reliable functional measure of walking ability.
Change in disease progression in SCA1 and SCA3 as determined by change in Cerebellar Cognitive Affective Syndrome (CCAS) score over time. | Every 12 months for approximately 60 months
  Cerebellar Cognitive Affective Syndrome Scale (CCAS Scale) is a battery of cognitive tasks used for determining the role of the cerebellum in the regulation of cognitive functions and present the procedure of neuropsychological diagnosis useful in indicating the specific cognitive and emotional problems in patients with cerebellar damage.
Change in disease progression in SCA1 and SCA3 as determined by change in Inventory of Non-ataxia Symptoms (INAS) total count over time. | Every 12 months for approximately 60 months
  Inventory of Non-ataxia Symptoms (INAS) is a scale utilized in recording the occurrence of accompanying non-ataxia symptoms. In the SARA validation trials, INAS was applied to a large number of SCA patients. Statistical evaluation showed good reliability.
Change in disease progression in SCA1 and SCA3 as determined by change in Functional staging score over time. | Every 12 months for approximately 60 months
  Functional staging is an instrument used to assess ambulatory capabilities of patients with cerebellar symptoms.
Change in level of disease activity based on change in cerebellar and brainstem volumes since baseline imaging. (Aim 2) | Every 12 months for approximately 36 months
  Change in level of disease activity based on change in cerebellar and brainstem volumes since baseline imaging.
Change in level of disease activity based on grey matter (GM) and white matter (WM) loss metrics from voxel-based morphometric (VBM) since baseline imaging. (Aim 2) | Every 12 months for approximately 36 months
  Change in level of disease activity as defined by change in grey matter volume and white matter volume from voxel-based morphometric data since baseline imaging.
Change in level of disease activity based on change in metabolite concentrations since baseline imaging. (Aim 2) | Every 12 months for approximately 36 months
  Change in level of disease activity on MR morphological, biochemical (MRS) and functional (resting-state fMRI) as defined by change in metabolite concentrations since baseline imaging.
Change in level of disease activity based on change in fractional isotropy since baseline imaging. (Aim 2) | Every 12 months for approximately 36 months
  Change in level of disease activity on MR morphological, biochemical (MRS) and functional (resting-state fMRI) as defined by change in mean diffusivity since baseline imaging.
Change in level of disease activity based on change in mean diffusivity since baseline imaging. (Aim 2) | Every 12 months for approximately 36 months
  Change in level of disease activity on MR morphological, biochemical (MRS) and functional (resting-state fMRI) as defined by change in mean diffusivity since baseline imaging.
Change in level of disease activity based on change in radial and axial diffusivity since baseline imaging. (Aim 2) | Every 12 months for approximately 36 months
  Change in level of disease activity on MR morphological, biochemical (MRS) and functional (resting-state fMRI) as defined by change in radial and axial diffusivity since baseline imaging.
Change in level of disease activity based on change in degree of co-activation within resting state networks since baseline imaging. (Aim 2) | Every 12 months for approximately 36 months
  Change in level of disease activity on MR morphological, biochemical (MRS) and functional (resting-state fMRI) as defined by change in degree of co-activation within resting state network since baseline imaging.

SECONDARY OUTCOMES:
Change in disease progression in SCA1 and SCA3 as determined by change in Friedreich's Ataxia Activities of Daily Living (FAA-ADL) over time. | Every 12 months for approximately 60 months
  Friedreich's Ataxia Activities of Daily Living (FAA-ADL) is an instrument measuring patient reported activities of daily living such as speech, dressing, walking, etc. Activities of daily living can be scored from 0-4, with zero being normal and 4 being most severe.
Change in disease progression in SCA1 and SCA3 as determined by change in Fatigue Severity Scale (FSS) over time. | Every 12 months for approximately 60 months
  Fatigue Severity Scale (FSS) is a 9 item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Scale ranges from 1-7, where 1 indicates strongly disagree and 7 indicates strongly agree.
Change in disease progression in SCA1 and SCA3 as determined by change in Euro Qol-5D (EQ-5D) over time. | Every 12 months for approximately 60 months
  Euro Qol-5D (EQ-5D), a measure developed by the EuroQol Group that generates a single index value for health status with considerable potential for use in health care evaluation.
Change in disease progression in SCA1 and SCA3 as determined by change in Patient Health Questionnaire (PHQ-9) over time. | Every 12 months for approximately 60 months
  Patient Health Questionnaire (PHQ-9) is a 9-question instrument used to screen for depression. The total of all 9 responses from the PHQ-9 aims to predict the presence and severity of depression.
Change in disease progression in SCA1 and SCA3 as determined by change in Patient Global Impression (PGI) over time. | Every 12 months for approximately 60 months
  Patient Global Impression (PGI) is patient reported measure of change in disease status, walking, hand function and speech since last visit or in the last 6 months. Changes can be reported as worse, stable/same, or improved/better.
Change in survival at 60 months between and within cohorts | Baseline to 60 months
  To compare survival of patients between and within cohorts at 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuo Ashizawa, MD, Study Chair — The Methodist Hospital Research Institute; Hank Paulson, MD, PhD, Study Director — University of Michigan; Gulin Oz, MD, Study Director — University of Minnesota; Thomas Klockgether, MD, Study Director — University Hospital Bonn - DZNE; Alexandra Durr, MD, PhD, Study Director — Hôpital Universitaire Pitié-Salpêtrière - ICM/SPATAX; Sheng Han Kuo, MD, Principal Investigator — Columbia University; George Wilmot, MD, PhD, Principal Investigator — Emory University; Liana Rosenthal, MD, Principal Investigator — Johns Hopkins University; Chiadikaobi Onyike, MD, Principal Investigator — Johns Hopkins University; Puneet Opal, MD, PhD, Principal Investigator — Northwestern University; Sharon Sha, Principal Investigator — Stanford University; Talene Yacoubian, MD, PhD, Principal Investigator — University of Alabama at Birmingham; Susan Perlman, MD, Principal Investigator — University of California, Los Angeles; Michael Geschwind, MD,PhD, Principal Investigator — University of California, San Francisco; Trevor Hawkins, MD, Principal Investigator — University of Colorado, Denver; Christopher Gomez, MD, PhD, Principal Investigator — University of Chicago; SH Subramony, MD, Principal Investigator — University of Florida; Vikram Shakkottai, MD, PhD, Principal Investigator — University of Texas; Khalaf Bushara, MD, Principal Investigator — University of Minnesota; Theresa Zesiewicz, MD, Principal Investigator — University of South Florida; Stefan Pulst, MD, PhD, Principal Investigator — University of Utah; Jeremy Schmahmann, MD, PhD, Principal Investigator — Harvard University; Peter Barker, MD, Principal Investigator — Johns Hopkins University; Haris I Sair, MD, Principal Investigator — Johns Hopkins University; Veronica Santini, MD, Principal Investigator — Stanford University; Eva-Maria Ratai, MD, Principal Investigator — Harvard University; Thomas Mareci, MD, Principal Investigator — Universtiy of Florida, Gainesville; Laura Scorr, MD, Principal Investigator — Emory University; Peggy C Nopoulos, MD, Principal Investigator — University of Iowa; Ali G Hamedani, MD, PhD, Principal Investigator — University of Pennsylvania; Yaz Y Kisanuki, MD, FAAN, Principal Investigator — Ohio State University; Peter Morrison, DO, Principal Investigator — University of Rochester
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paulson HL, Shakkottai VG, Clark HB, Orr HT. Polyglutamine spinocerebellar ataxias - from genes to potential treatments. Nat Rev Neurosci. 2017 Oct;18(10):613-626. doi: 10.1038/nrn.2017.92. Epub 2017 Aug 17. PMID 28855740
- [Background] Ashizawa T, Figueroa KP, Perlman SL, Gomez CM, Wilmot GR, Schmahmann JD, Ying SH, Zesiewicz TA, Paulson HL, Shakkottai VG, Bushara KO, Kuo SH, Geschwind MD, Xia G, Mazzoni P, Krischer JP, Cuthbertson D, Holbert AR, Ferguson JH, Pulst SM, Subramony SH. Clinical characteristics of patients with spinocerebellar ataxias 1, 2, 3 and 6 in the US; a prospective observational study. Orphanet J Rare Dis. 2013 Nov 13;8:177. doi: 10.1186/1750-1172-8-177. PMID 24225362
- [Background] Oz G, Hutter D, Tkac I, Clark HB, Gross MD, Jiang H, Eberly LE, Bushara KO, Gomez CM. Neurochemical alterations in spinocerebellar ataxia type 1 and their correlations with clinical status. Mov Disord. 2010 Jul 15;25(9):1253-61. doi: 10.1002/mds.23067. PMID 20310029
- [Background] Tezenas du Montcel S, Durr A, Rakowicz M, Nanetti L, Charles P, Sulek A, Mariotti C, Rola R, Schols L, Bauer P, Dufaure-Gare I, Jacobi H, Forlani S, Schmitz-Hubsch T, Filla A, Timmann D, van de Warrenburg BP, Marelli C, Kang JS, Giunti P, Cook A, Baliko L, Melegh B, Boesch S, Szymanski S, Berciano J, Infante J, Buerk K, Masciullo M, Di Fabio R, Depondt C, Ratka S, Stevanin G, Klockgether T, Brice A, Golmard JL. Prediction of the age at onset in spinocerebellar ataxia type 1, 2, 3 and 6. J Med Genet. 2014 Jul;51(7):479-86. doi: 10.1136/jmedgenet-2013-102200. Epub 2014 Apr 29. PMID 24780882
- [Derived] Arpin DJ, Subramony SH; READISCA Consortium; Vaillancourt DE, Ashizawa T, Durr A, Mareci T, Klockgether T, Faber J, Paulson HL, Oz G, Burns MR. Fixel-Based Analysis of Diffusion Imaging as a Quantitative Marker of Disease State in Spinocerebellar Ataxia. Ann Clin Transl Neurol. 2025 Sep;12(9):1846-1857. doi: 10.1002/acn3.70116. Epub 2025 Jul 15. PMID 40665587
- [Derived] Tezenas du Montcel S, Petit E, Olubajo T, Faber J, Lallemant-Dudek P, Bushara K, Perlman S, Subramony SH, Morgan D, Jackman B, Figueroa KP, Pulst SM, Fauret-Amsellem AL, Dufke C, Paulson HL, Oz G, Klockgether T, Durr A, Ashizawa T; READISCA Consortium Collaborators. Baseline Clinical and Blood Biomarkers in Patients With Preataxic and Early-Stage Disease Spinocerebellar Ataxia 1 and 3. Neurology. 2023 Apr 25;100(17):e1836-e1848. doi: 10.1212/WNL.0000000000207088. Epub 2023 Feb 16. PMID 36797067